CLINICAL TRIAL: NCT00005893
Title: Study of Allogeneic Bone Marrow Transplantation Using Matched, Related Donors in Patients With Nonmalignant Hematologic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fairview University Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15101; UMN-MT-1994-18; UMN-MT-9418
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Neutropenia; Sickle Cell Anemia; Thalassemia Major; Red-Cell Aplasia, Pure
Keywords: chronic congenital neutropenia; chronic neutropenia; congenital pure red cell aplasia; disease-related problem/condition; genetic diseases and dysmorphic syndromes; hematologic disorders; neutropenia; pure red cell aplasia; rare disease; sickle cell anemia; thalassemia major
MeSH Terms: conditions — Neutropenia; Anemia, Sickle Cell; beta-Thalassemia; Red-Cell Aplasia, Pure; Anemia, Diamond-Blackfan; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Bone Marrow Transplantation

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Procedure: Bone marrow transplantation

SUMMARY:
OBJECTIVES: I. Determine the efficacy of bone marrow transplantation using matched related donors in patients with nonmalignant hematologic disorders.

II. Determine the quality of life, absence of adverse effects (e.g., graft versus host disease and B cell lymphoproliferative disease), and completeness of recovery of their underlying condition in these patients with this treatment regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive IV or oral busulfan every 6 hours on days -9 to -6; cyclophosphamide IV on days -5 to -2; anti-thymocyte globulin IV on days -4 to -2; and allogeneic bone marrow transplantation (BMT) on day 0.

Patients with class 3 thalassemia (liver edge greater than 2 cm below costal margin, a history of inconsistent chelation, and portal fibrosis) receive a less intensive conditioning regimen consisting of oral busulfan every 6 hours on days -7 to -4; anti-thymocyte globulin IV on days -5 to -1 and days 1-5; cyclophosphamide IV on days -3 to -2; and allogeneic BMT on day 0.

Patients are followed at day 28, and then at 3, 6, 12, and 24 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Severe hemoglobinopathy including, but not limited to the following:

Homozygous beta thalassemia Other beta chain mutation as demonstrated by hemoglobin electrophoresis Sickle cell anemia (age 16 to 50 years) Evidence of one or more the following prior complications: Stage I-II sickle cell lung disease Sickle cell nephropathy (moderate to severe proteinuria or glomerular filtration rate of 30-50% predicted normal for age) Acute chest syndrome requiring blood transfusions More than 3 debilitating pain episodes per year for 3 years lasting more than 4 hours each Any combination of episodes of acute chest syndrome and painful episodes adding up to 3 episodes per year for 3 consecutive years Requirement for chronic transfusions with alloimmunization (more than 2 antibodies) Sickle cell anemia (age under 16 years) Evidence of one or more the following prior complications: Prior stroke or hemorrhage Any neurologic event lasting more than 24 hours Abnormal cerebral MRI and cerebral arteriogram MRI angiographic impaired neuropsychologic testing Stage I-II sickle cell lung disease Sickle cell nephropathy (moderate to severe proteinuria or glomerular filtration rate of 30-50% predicted normal for age) Significant visual impairment in at least one eye with bilateral proliferative retinopathy Acute chest syndrome with history of recurrent hospitalizations or exchange transfusions Osteonecrosis of multiple joints with destructive changes More than 3 debilitating pain episodes per year or priapism Requirement for chronic transfusions with alloimmunization

OR

Bone marrow failure syndrome unresponsive to therapy, including but not limited to the following: Congenital pure red cell aplasia (Diamond Blackfan anemia) Confirmed by bone marrow aspirate More than 6 transfusions per year despite steroid therapy Kostmann's neutropenia Confirmed by bone marrow aspirate Unable to maintain absolute neutrophil count greater than 750/mm3 or recurrent life threatening infections or more than 4 hospitalizations per year despite therapy with filgrastim (G-CSF) No myelodysplasia or aplastic anemia

Must have a related donor with at least a 5 out of 6 HLA antigen match

--Patient Characteristics--

Age: Sickle cell anemia patients 0 to 50; All other patients under 18

Performance status: Karnofsky 70-100%

Hepatic: Bilirubin no greater than 3.0 mg/dL with a direct fraction no greater than 2.0 mg/dL ALT no greater than 150 U/L No moderate or severe portal fibrosis No active hepatitis

Renal: Glomerular filtration rate at least 30% predicted (except with sickle cell anemia) No renal dysfunction

Cardiovascular: Left ejection fraction at least 50% No cardiac compromise

Other: No severe, stable neurologic impairment HIV negative

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Orchard, Study Chair — Fairview University Medical Center
Locations (1):
- Fairview University Medical Center, Minneapolis, Minnesota, United States